CLINICAL TRIAL: NCT01964625
Title: Assessment of Positron Emission Tomography - Computed Tomography (PET-CT) Scanning as a Potential Biomarker to Assess Disease Activity in Chronic Graft Versus Host Disease (GvHD): A Pilot Study
Brief Title: Positron Emission Tomography - Computed Tomography (PET-CT) Scanning in Chronic Graft Versus Host Disease (cGvHD)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated due to lack of enrollment
Sponsor: University of Rochester (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 32186
Record Dates: First submitted 2010-12-01; First posted 2013-10-17 (Estimated); Last update posted 2013-10-17 (Estimated); Status verified 2013-10

CONDITIONS: Chronic Graft Versus Host Disease
Keywords: Chronic GvHD
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PET-CT (Experimental): Patients who have a negative routine PET-CT evaluation followed by onset and confirmation in accordance with NIH guidelines, will receive another PET-CT scan prior to initiation of therapy for chronic GvHD.
  Interventions: Other: PET-CT Scan

INTERVENTIONS:
Other: PET-CT Scan — PET-CT scan will be done at baseline (per standard of care), at onset and confirmation of chronic GvHD and after initiation of therapy to assess response.

SUMMARY:
Graft versus Host Disease (GvHD), in both its acute and chronic forms, is the major intrinsic complication of allogeneic hematopoeitic stem cell transplant (allo-HSCT). Moreover, chronic GvHD may be regarded as a "late effect" of cancer therapy, and the severity of chronic GvHD is the chief determinant of long-term survival following allo-HSCT. Unfortunately, the investigators understanding (and thus management) of chronic GvHD is not optimal; a recent NIH Consensus Conference has defined inadequacies in virtually all facets of chronic GvHD management. Notably for this study, the lack of suitable biomarkers compromises diagnosis, staging and therapeutic response evaluation of chronic GvHD - and also hinders better understanding of the biology of this process.

In particular, the activity of chronic GvHD is often difficult to discern, potentially causing either undertreatment, with the risk of morbidity and/or mortality due to uncontrolled chronic GvHD, or possibly overtreatment, with potent ISTs causing unnecessary toxicity. Obviously, the development of reliable biomarkers of chronic GvHD activity would be a very useful advance in addressing this problem, as well as other facets of management not addressed due to certain limitations, as detailed herein.

Potentially, certain imaging technologies could address this problem. To date, imaging technology has been used only sporadically in chronic GvHD and is not an integral part of routine assessments. However, and despite its nonspecific nature, certain "inflammatory" features of some chronic GvHD cases, plus clinical similarity to certain autoimmune diseases in which functional imaging has been tested in research trials - (and perhaps notably), a limited experience in acute GvHD - the investigators postulate that Positron emission tomography - computed tomography (PET-CT) scans may be useful as a biomarker of disease activity in chronic GvHD. This protocol is an initial effort to that end.

ELIGIBILITY:
Inclusion Criteria:

* Prior allogeneic hematopoietic stem cell transplant (+/- DLI)
* As per current recommendations, no interval from allo HSCT will be required to differentiate acute from chronic Graft versus Host Disease (GvHD)
* Patients must have had negative routine restaging PET-CT scans
* Patients may not have had any more than two weeks' specific treatment for chronic GvHD. (It is recognized that some patients develop chronic GvHD while on immunosuppressive prophylaxis; such patients will remain eligible, even if dose adjustment of these prophylactic agents occurs. The "two week" interval pertains to the use of additional agents in this case.)
* Diagnosis of chronic GvHD must be confirmed. In the usual case, tissue biopsy will be required; however, some chronic GvHD patients do not require tissue biopsy for confirmation. The PI and co-investigator must agree on eligibility.
* Per patient approval by PI and one additional co-investigator
* Informed consent

Exclusion Criteria:

* Patients with a malignancy not in remission will be excluded.
* Negative routine pregnancy testing. Patients either pregnant or unwilling to use satisfactory contraception (if appropriate) will not be eligible. All female patients must use a highly effective birth control method or a combination of 2 additionally effective birth control methods while in this study. Examples of highly effective birth control are: a condom or a diaphragm with spermicidal jelly, oral, injectable, or implanted birth control, or abstinence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2010-11; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
To determine ability of PET-CT scans to delineate and stage initial chronic GvHD | At initial diagnosis of chronic GvHD
  Assessment to take place after confirmed diagnosis of chronic GvHD but before initiation of therapy

SECONDARY OUTCOMES:
To determine ability of PET-CT scans to document response to chronic GvHD therapy | PET-CT performed </= 6 months from study PET-CT #1
  Therapy for chronic GvHD can be standard of care or investigational. Maximal response to treatment is defined as stability on two occasions >/= one month apart; PET-CT to be performed within two weeks of this assessment. Initial PET-CT at diagnosis will be used as the comparison.

CONTACTS AND LOCATIONS:
Overall Officials: Gordon L Phillips, II, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States